CLINICAL TRIAL: NCT06097585
Title: Effect of Gliflozins on Heart Failure Due to Regurgitant Rheumatic Valve Disease
Brief Title: Gliflozins on HF in Regurgitant Rheumatic Heart
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Youssef Dandrawy, residant doctor, Assiut University
Other Study IDs: gliflozins on rheumatic HF
Record Dates: First submitted 2023-09-30; First posted 2023-10-24 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Rheumatic Heart Disease; Heart Failure
MeSH Terms: conditions — Rheumatic Heart Disease; Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SGLT2I Group: the case group that will receive SGLT2I in the treatment
  Interventions: Drug: SGLT2 inhibitor
- non - SGLT2I Group: the control group that will not receive SGLT2I in the treatment

INTERVENTIONS:
Drug: SGLT2 inhibitor — case control study in which group will receive SGLT2I and group will not , to detect impact of the drug in changing NYHA class for heart failure and echographic parameter
  Other Names: gliflozins
  Groups: SGLT2I Group

SUMMARY:
The objective of this trial is to detect impact of Gliflozin on patients with heart failure due to reurgitant rheumatic valve disease

DETAILED DESCRIPTION:
* Rheumatic heart disease is a chronic sequel of acute rheumatic fever caused by group A β hemolytic Streptococcal pharyngitis and possibly pyoderma, which mimics molecular heart structures so the immune response leads to carditis and valvular heart damage. Damage to valves cause mitral and/or aortic regurgitation, or in long-standing stenosis. Complications of rheumatic heart disease include heart failure, embolic stroke, endocarditis and atrial fibrillation .
* Heart failure (HF) is a progressive syndrome characterised by the inability of the heart to provide adequate blood supply to meet the metabolic demand of different tissues .
* The recent ESC/AHA/ACC guidelines of HF set medications as class 1 for the HF therapy as ACE-I/ ARNI/beta-blocker/MRA/ SGLT2 I as they reduced the risk of cardiovascular death and worsening HF in patients with HFrEF , Unless contraindicated or not tolerated.
* Empagliflozin is an orally available inhibitor sodium glucose co-transporter 2 receptor (SGLT-2), empagliflozin exerts its effect by preventing sodium and glucose reabsorption from proximal convoluted tubules. This leads to increased urinary sodium and glucose excretion, This is associated with a modest osmotic diuresis, blood pressure lowering effect, improvement in arterial stiffness , and decrease in heart rate.
* DAPA-HF trial shows: The primary outcome of cardiovascular death, HF hospitalization, for dapagliflozin vs. placebo, was 16.3% vs 21.2% (p < 0.001).
* EMPA-REG OUTCOME trial shows: The primary outcome, cardiovascular death or HF hospitalization, for empagliflozin vs. placebo, was 19.4% vs. 24.7% ( p < 0.001).

ELIGIBILITY:
Inclusion Criteria:

* All male or female patients having rheumatic heart disease with either mitral, aortic, tricuspid regurge as a single or combined valvular lesion
* Patients aged 18 years or older at time of inclusion in the study
* Patients with HF currently in NYHA class II-IV, or asymptomatic patients with proved mitral regurgitant lesion.
* Body Mass Index (BMI) < 45 kg/m2

Exclusion Criteria:

* Advanced stage liver and kidney failure (glomerular filtration rate < 20 mL/min/1.73 m2).
* Patient with implanted cardiac pacemaker, implantable cardioverter-defibrillator (ICD) or cardiac re-synchronization therapy (CRT) or implanted left ventricular assist device (LVAD)
* Diagnosis of cardiomyopathy induced by other etiologies rather than rheumatic heart disease eg, ischemia , dilated cardiomyopathy,…..etc within the 12 months prior to Visit 1
* Known allergy or hypersensitivity to SGLT-2 inhibitors
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* ongoing hematological diseases and malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending outpatient clinic, cardiology department, Assiut university hospital and south valley university hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of the clinical condition | 6 months up to 1 year
  improving or worsening in NYHA class: I- Ordinary physical activity does not cause undue fatigue, dyspnea, or palpitations.
  II- Ordinary physical activity causes fatigue, dyspnea, palpitations, or angina.
  III- Comfortable at rest; less than ordinary physical activity causes fatigue, dyspnea, palpitations, or angina.
  IV- Symptoms occur at rest; any physical activity increases discomfort.
change of the function and regurge | 6 months up to 1 year
  improving or worsening in echocardiographic parameter :
  * ejection fraction by simpson methods
  * severity of regurge by color Doppler and continuous wave Doppler

SECONDARY OUTCOMES:
major adverse cardiovascular event | 6 months up to 1 year
  monitor rate for Cardiovascular death, non-fatal stroke, non-fatal myocardial infarction and hospitalization for HF between 2 groups
Glomerular filtration rate affection | 6 months up to 1 year
  monitor rate of decline in the estimated glomerular filtration rate between 2 groups
urinary tract infection | 6 months up to 1 year
  incidence of urinary tract infection between 2 groups by following urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Fouad, MD, Study Director — Assiut University; Magdy A Algowhary, MD, Study Director — Assiut University; Ahmed G Bakry, MD, Study Director — South Valley University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Background] Inzucchi SE, Zinman B, Wanner C, Ferrari R, Fitchett D, Hantel S, Espadero RM, Woerle HJ, Broedl UC, Johansen OE. SGLT-2 inhibitors and cardiovascular risk: proposed pathways and review of ongoing outcome trials. Diab Vasc Dis Res. 2015 Mar;12(2):90-100. doi: 10.1177/1479164114559852. Epub 2015 Jan 14. PMID 25589482
- [Background] Chilton R, Tikkanen I, Cannon CP, Crowe S, Woerle HJ, Broedl UC, Johansen OE. Effects of empagliflozin on blood pressure and markers of arterial stiffness and vascular resistance in patients with type 2 diabetes. Diabetes Obes Metab. 2015 Dec;17(12):1180-93. doi: 10.1111/dom.12572. Epub 2015 Oct 9. PMID 26343814
- [Background] Fitchett D, Inzucchi SE, Cannon CP, McGuire DK, Scirica BM, Johansen OE, Sambevski S, Kaspers S, Pfarr E, George JT, Zinman B. Empagliflozin Reduced Mortality and Hospitalization for Heart Failure Across the Spectrum of Cardiovascular Risk in the EMPA-REG OUTCOME Trial. Circulation. 2019 Mar 12;139(11):1384-1395. doi: 10.1161/CIRCULATIONAHA.118.037778. PMID 30586757
- [Background] Zuhlke LJ, Beaton A, Engel ME, Hugo-Hamman CT, Karthikeyan G, Katzenellenbogen JM, Ntusi N, Ralph AP, Saxena A, Smeesters PR, Watkins D, Zilla P, Carapetis J. Group A Streptococcus, Acute Rheumatic Fever and Rheumatic Heart Disease: Epidemiology and Clinical Considerations. Curr Treat Options Cardiovasc Med. 2017 Feb;19(2):15. doi: 10.1007/s11936-017-0513-y. PMID 28285457
- [Background] Carapetis JR, Beaton A, Cunningham MW, Guilherme L, Karthikeyan G, Mayosi BM, Sable C, Steer A, Wilson N, Wyber R, Zuhlke L. Acute rheumatic fever and rheumatic heart disease. Nat Rev Dis Primers. 2016 Jan 14;2:15084. doi: 10.1038/nrdp.2015.84. PMID 27188830
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829